CLINICAL TRIAL: NCT05122078
Title: Effects of Analgesia Nociception Index (ANI)-Guided Analgesia on Postoperative Bowel Function Recovery in Laparoscopic Colorectal Surgery: A Prospective Randomized-controlled Study
Brief Title: Effects of Analgesia Nociception Index (ANI)-Guided Analgesia on Postoperative Bowel Function.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Young Song, Associate Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3-2021-0348
Record Dates: First submitted 2021-11-04; First posted 2021-11-16 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Postoperative Bowel Function Recovery
Keywords: Analgesia Nociception Index (ANI)

STUDY DESIGN:
Intervention Model Description: Single blinded randomized controlled study
Who Masked: Participant
Masking Description: Patients don't know which group they belong to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ANI group (Experimental): Investigator will attach the ANI monitor V2 (MDoloris Medical Systems, Lille, France) to the patient and monitor Analgesia Nociception Index (ANI) during anesthesia. Remifentanil infusion rate is adjusted according to ANI monitoring. The ANI is adjusted to be between 50 and 70.
  Interventions: Device: ANI; Other: Control
- Control group (No Intervention): Remifentanil infusion rate is adjusted according to the conventional method of blood pressure and heart rate monitroing. Blood pressure and heart rate are controlled to be within 20% of baseline. We will not monitor ANI in this group.

INTERVENTIONS:
Device: ANI — Investigators will attach the ANI monitor V2 (MDoloris Medical Systems, Lille, France) to the patient and monitor Analgesia Nociception Index (ANI) during anesthesia. Remifentanil infusion rate is adjusted according to ANI monitoring. The ANI is adjusted to be between 50 and 70.
  Arms: ANI group
Other: Control — Remifentanil infusion rate is adjusted according to the conventional method of blood pressure and heart rate monitroing. Blood pressure and heart rate are controlled to be within 20% of baseline. Investigators will not monitor ANI in this group.
  Arms: ANI group

SUMMARY:
Investigators will examaine the effects of Analgesia Nociception Index (ANI)-guided analgesia on postoperative bowel function recovery in laparoscopic colorectal surgery. This is a prospective randomized-controlled study.

Investigators will randomly divide the patients into two groups. In ANI group, remifentanil infusion rate during anesthesia will be adjusted according to ANI monitoring. In Control group, remifentanil infusion rate during anesthesia will be adjusted according to the conventional method of blood pressure and heart rate monitroing. And Investigators will evalualte the bowel function recovery in both groups after surgery, and compare between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 19 years who undergo laparoscopic colorectal surgery for colorectal cancer at Gangnam Severance Hospital, Seoul, South Korea.

Exclusion Criteria:

* Emergency surgery
* Patients with history of open abdominal surgery
* Patients with arrhythmia
* Patients with pacemaker insertion
* Patients with history of heart transplantation
* Patients taking medications that may affect ANI (antimuscarinics, alpha-agonists, beta blockers)
* Patients with chronic opioid medication.
* Cognitive impairment
* Unable to read consent form (eg illiterate, foreigner, etc.)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2025-10-14 (Estimated); Study Completion 2025-10-14 (Estimated)

PRIMARY OUTCOMES:
Time to first gas passing from surgery | Up to postoperative 2weeks
  Time (hours) to first gas passing from surgery

SECONDARY OUTCOMES:
Time to starting fluid intake from surgery | up to 2weeks
  Time (hours) to starting oral fluid intake after surgery
Time to starting soft diet from surgery | up to 2 weeks
  Time (hours) to starting soft diet from surgery
Intraoperative opioid consumption | during anesthesia
  Total opioid dose administered to the patient during anesthesia
Postoperative opioid consumption | postoperative 6hours, 12hours, 24hours, 36hours, 48hours, 3days, 4days, 5days.(Minimum value: 0, Maximum value: 10, higher score means worse.)
  Total opioid dose administered to the patient after surgery.
Pain score | postoperative 6hours, 12hours, 24hours, 36hours, 48hours, 3days, 4days, 5days.(Minimum value: 0, Maximum value: 10, higher score means worse.)
  Visual analog scale (VAS) 0-10
Nausea score | postoperative 6hours, 12hours, 24hours, 36hours, 48hours, 3days, 4days, 5days
  verbal numerical rating scale 0-10
Time to first rescue analgesics from surgery | up to 2weeks
  Time (hours) to first rescue analgesics from surgery.
Number of vomiting, antiemetic administration | up to 2weeks
  Number of vomiting, antiemetic administration
Time to starting ambulation from surgery. | up to 2 weeks
  Time (hours) to starting ambulation from surgery
QoR-15 | postoperative 1days, 4days
  Score of QoR-15 questionnaire (Quality of Recovery-15) (Minimum value: 0, Maximum value: 150, higher score means better.)
Hemodynamics during anesthesia | during anesthesia
  hemodynamics (blood pressure, heart rate) during anesthesia
Plasma concentration of Cortisol, Norepinephrine, Epinephrine, IL-6 | immediately after surgery
  Plasma concentration of Cortisol(mcg/dL), Norepinephrine(pg/mL), Epinephrine(pg/mL), IL-6(pg/mL) immediately after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- GangnamSeverance Hospital, Seoul, South Korea